CLINICAL TRIAL: NCT05521035
Title: Risk and Incidence of Aortic Graft and Endograft Infection in Patients With Bloodstream Infection, a Population Based Study in South Sweden
Brief Title: Risk and Incidence of Aortic Graft and Endograft Infection With BSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-5-BSI
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Aortic Infections and Inflammations
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is the risk of aortic vascular graft and endograft infection in patients with aortic vascular graft/endograft and bloodstream infection?

DETAILED DESCRIPTION:
All patients with previous aortic vascular graft and endograft surgery between years 2010 and 2021 in four regions of south Sweden (Skåne, Halland, Kronoberg and Blekinge) will be included in the study. These patients will be evaluated for bloodstream infection (BSI) or not. For all patients with BSI, the risk of aortic vascular graft and endograft infection will be investigated. Aortic vascular graft and endograft infection will be determined by usage of the MAGIC-criteria.

Risk factors for developing aortic vascular graft and endograft infection will be investigated, and if possible used to construct a risk score. This risk score could be used by clinicians to determine if bacteremic patients with aortic vascular grafts or endografts should be evaluated for aortic vascular graft and endograft infection.

ELIGIBILITY:
Inclusion Criteria:

Previous aortic vascular graft or endograft infection with bloodstream infection.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with previous aortic vascular graft or endograft surgery in Skåne, Halland, Kronoberg and Blekinge between the years 2010-2021.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Aortic vascular graft or endograft infection | At least 1 year follow-up
  Determined by the MAGIC-criteria

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ljungquist, Principal Investigator — Lund University
Locations (1):
- Helsingborgs lasarett, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
If individual participant data (IPD) will be shared, it will be after researchers has been given ethical approval

REFERENCES:
- See also: Treatment and outcomes of aortic endograft infection — https://pubmed.ncbi.nlm.nih.gov/26804214/
- See also: Diagnosis of Aortic Graft Infection: A Case Definition by the Management of Aortic Graft Infection Collaboration (MAGIC) — https://pubmed.ncbi.nlm.nih.gov/27771318/
- See also: Secondary infections of thoracic and abdominal aortic endografts — https://pubmed.ncbi.nlm.nih.gov/19097807/